CLINICAL TRIAL: NCT07032207
Title: The Correlation of Gastric Residual Volume Detected by Preoperative Gastric Ultrasonography With Body Mass Index and Aspiration Risk in Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Correlation of Preoperative Gastric Residual Volume With Body Mass Index and Aspiration Risk in Laparoscopic Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Büşra Tanacıoğlu, Research Assistant MD, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH-BT01
Record Dates: First submitted 2025-05-19; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Gastric Ultrasound; Gastric Residual Volume; Body Mass Index (BMI)
Keywords: obesity; gastric ultrasound; gastric residual volume; body mass index; aspiration
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is a chronic, complex disease defined by the World Health Organization (WHO) as the excessive accumulation of fat in the body that can harm health. Since 1975, the prevalence of obesity has been increasing worldwide, making it a significant public health issue. Body mass index (BMI) is important in diagnosing obesity. BMI is calculated by dividing a person's weight (kg) by the square of their height (m²). BMI: weight (kg) / height² (m²). According to the WHO, a BMI between 30.0-34.9 kg/m² is classified as Class 1 obesity, between 35.0-39.9 kg/m² as Class 2 obesity, between 40-49.9 kg/m² as Class 3 obesity, and ≥50.0 kg/m² as super obesity.

Obesity is closely related to increasing morbidity and mortality worldwide, and in obese patients, the incidence of diseases such as type 2 diabetes, hypertension, cardiovascular disease, dyslipidemia, coronary heart disease, obstructive sleep apnea, asthma, depression, other psychiatric disorders, and gastroesophageal reflux has increased. Treatment options for obesity include lifestyle changes, specific diets, diet-drug combinations, metabolic and various bariatric surgical options. Among these treatment options, metabolic and bariatric surgical procedures are considered the most effective methods for weight loss.

Aspiration of gastric contents is a significant perioperative complication that can cause up to 9% of anesthesia-related deaths. Due to delayed gastric emptying in obese patients, the risk of aspiration is higher compared to non-obese patients. In obese patients, preoperative anesthesia management is more challenging, and the risk of pulmonary aspiration is greater. Since obesity is an independent risk factor for patients with a full stomach, and airway management can be difficult in these patients, it is essential to assess the aspiration risk in the preoperative period.

Anesthesia guidelines recommend that to improve the quality and effectiveness of anesthesia care and reduce the severity of potential complications related to perioperative pulmonary aspiration of gastric contents, adults and children should be allowed to drink clear liquids up to 2 hours before elective surgery, and solid food consumption should be prohibited 6 hours before elective surgery.

Recently, with the integration of ultrasound into anesthesia practice, ultrasound has been applied in various surgical procedures and clinical conditions. The use of ultrasound to evaluate the risk of aspiration in the preoperative period and to determine the residual gastric volume is increasingly being used in clinical practice. The use of gastric ultrasound to assess aspiration risk has also been increasing in pediatric patient groups and pregnant patients, similar to obese patient groups.

In this study, the investigators' aim is to determine the relationship between BMI, fasting duration, and aspiration risk by assessing the gastric residual volume in the preoperative period through gastric ultrasonography in patients with obesity who will undergo bariatric surgery.

DETAILED DESCRIPTION:
Patients will be informed about the study procedure one day before the surgery, and informed consent will be obtained from those who agree to participate. For patients who have given consent, gastric ultrasonography will be performed in the anesthesia preparation room before surgery. The examination will be conducted first in the supine position and then in the right lateral decubitus (RLD) position.

While patients are in the RLD and supine positions, a low-frequency (2-5 MHz) curved ultrasound probe will be used to scan from left to right along the subcostal margin. The left lobe of the liver and the descending abdominal aorta will be used as anterior and posterior landmarks. Gastric content will be evaluated both qualitatively and quantitatively by gastric ultrasonography.

In the RLD position, two maximum perpendicular diameters of the stomach-anteroposterior (AP) and craniocaudal (CC)-will be measured. The antral cross-sectional area (CSA) in the right lateral decubitus position will be calculated using the formula:

CSA = (AP × CC × π) / 4.

Gastric residual volume will then be calculated using the formula by Perlas et al.:

Gastric residual volume (mL) = 27.0 + 14.6 × right lateral CSA - 1.28 × age.

Patients with an empty antrum and gastric residual volume less than 1.5 mL/kg will be considered at low risk for aspiration, whereas those with solid content and/or gastric residual volume greater than 1.5 mL/kg will be considered high risk for aspiration. A flat antrum image with anterior and posterior walls adjacent will be regarded as an empty stomach. A hypoechoic, thin-walled, distended antrum will be interpreted as liquid content, and a distended antrum showing mixed echogenicity on ultrasound will be considered solid content.

Additionally, the antrum will be classified using a three-point grading system:

Grade 0: No fluid visible in both supine and RLD positions.

Grade 1: Clear fluid visible only in the RLD position.

Grade 2: Fluid and solid content visible in both supine and RLD positions.

All measurements will be repeated three times, and the average will be taken. The duration of the ultrasonography procedure will be recorded.

Preoperative laboratory values including fasting blood glucose, HbA1c, renal function tests (urea, creatinine), liver function tests (AST, ALT), serum electrolytes (sodium, potassium, chloride, calcium), hemogram parameters (hemoglobin, hematocrit, platelet, leukocyte), and coagulation parameters (APTT, INR) will be documented.

Demographic data (age, gender, height, weight), BMI, waist circumference, xiphoid circumference, ASA score, comorbidities, previous surgeries, and ongoing medications will also be recorded.

After completing the gastric ultrasonography, patients will be taken to the operating room. Standard monitoring including electrocardiogram (ECG), non-invasive blood pressure, peripheral oxygen saturation (SpO2), and bispectral index (BIS) will be applied. Premedication will be performed with intravenous midazolam 0.02 mg/kg, followed by preoxygenation with 100% oxygen via mask for 3 minutes.

Standard anesthesia induction will be carried out using intravenous propofol 2-2.5 mg/kg, fentanyl 2 mcg/kg, and rocuronium 0.6 mg/kg. Orotracheal intubation will be performed once adequate muscle relaxation is achieved. Mechanical ventilation will be provided in volume control mode with tidal volumes of 6-8 ml/kg and end-tidal carbon dioxide (EtCO2) maintained between 35-40 mmHg.

Anesthesia maintenance will be ensured with sevoflurane 1.5-2% in 2 L/min of 50% oxygen-air mixture and intravenous remifentanil infusion at 0.05-0.5 mcg/kg/min, targeting BIS values between 40-60. Normothermia will be maintained intraoperatively with active forced-air warming devices in all patients.

Perioperative aspiration events will be recorded as "occurred" or "not occurred." Total surgical and anesthesia durations will be documented.

Twenty minutes before the end of surgery, patients will receive postoperative analgesia prophylaxis with intravenous administration of 1 g paracetamol, 1 mg/kg tramadol, and 4 mg ondansetron for nausea and vomiting prophylaxis, according to our standard protocol.

At the end of surgery, anesthetic agents will be discontinued, and the awakening phase will begin. After patients resume spontaneous respiration, neuromuscular blockade will be reversed with intravenous sugammadex 2 mg/kg. Patients with adequate respiratory effort and BIS ≥ 85 will be extubated and transferred to the recovery unit once they are awake, have regained muscle strength, and are hemodynamically stable.

Postoperative nausea will be evaluated at 1, 6, and 24 hours using a 5-point nausea-vomiting severity scale (0 = no nausea, 1 = mild nausea without vomiting, 2 = moderate nausea with vomiting, 3 = vomiting less than twice per hour, 4 = vomiting more than twice per hour) and any complications will be recorded (present/absent).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo bariatric surgery under general anesthesia in elective conditions
* Patients in ASA II-III groups, with BMI > 35 kg/m², and aged between 18-65 years
* Patients who have provided informed consent

Exclusion Criteria:

* Patients under 18 years of age, over 65 years of age, or in ASA IV-V groups
* Pregnancy
* Patients with upper gastrointestinal (GI) abnormalities such as hiatal hernia and gastric tumors
* Patients with a recent history of upper GI bleeding (within the last 12 months), previous stomach and esophagus surgeries, or abnormal anatomy of the upper gastrointestinal tract
* Patients using medications that affect gastric motility or other related conditions
* Patients with uncontrolled diabetes
* Patients who require emergency surgery
* Patients with advanced cardiac, renal, pulmonary, or hepatic failure
* Patients who refuse to participate and do not provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo bariatric surgery under general anesthesia in elective conditions
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The correlation between BMI, gastric residual volume, and aspiration risk. | 5 minutes
  Higher BMI levels may be associated with increased gastric residual volume (GRV), which in turn can elevate the risk of pulmonary aspiration, especially during anesthesia. Understanding the correlation between BMI, GRV, and aspiration risk is crucial for developing safer preoperative fasting guidelines and optimizing care in high-risk patients.

SECONDARY OUTCOMES:
The correlation between fasting duration, gastric residual volume, and the risk of aspiration | 5 minutes
  Understanding this correlation is crucial in clinical settings, especially in anesthesia, as prolonged fasting may not always reduce gastric volume or aspiration risk. The goal is to optimize preoperative fasting time to enhance patient safety and comfort while minimizing complications related to aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU YILDIRIM AR, Associate Professor, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherwin M, Katz D. Using gastric ultrasound to assess gastric content in the pregnant patient. BJA Educ. 2021 Nov;21(11):404-407. doi: 10.1016/j.bjae.2021.08.001. Epub 2021 Sep 23. No abstract available. PMID 34707884
- [Background] Moake MM, Presley BC, Hill JG, Wolf BJ, Kane ID, Busch CE, Jackson BF. Point-of-Care Ultrasound to Assess Gastric Content in Pediatric Emergency Department Procedural Sedation Patients. Pediatr Emerg Care. 2022 Jan 1;38(1):e178-e186. doi: 10.1097/PEC.0000000000002198. PMID 32769837
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Bouvet L, Desgranges FP, Aubergy C, Boselli E, Dupont G, Allaouchiche B, Chassard D. Prevalence and factors predictive of full stomach in elective and emergency surgical patients: a prospective cohort study. Br J Anaesth. 2017 Mar 1;118(3):372-379. doi: 10.1093/bja/aew462. PMID 28203726
- [Background] Mahajan V, Hashmi J, Singh R, Samra T, Aneja S. Comparative evaluation of gastric pH and volume in morbidly obese and lean patients undergoing elective surgery and effect of aspiration prophylaxis. J Clin Anesth. 2015 Aug;27(5):396-400. doi: 10.1016/j.jclinane.2015.03.004. Epub 2015 Apr 30. PMID 25935831
- [Background] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Background] Singhal V, Youssef S, Misra M. Use of sleeve gastrectomy in adolescents and young adults with severe obesity. Curr Opin Pediatr. 2020 Aug;32(4):547-553. doi: 10.1097/MOP.0000000000000927. PMID 32692052
- [Background] Aaseth J, Ellefsen S, Alehagen U, Sundfor TM, Alexander J. Diets and drugs for weight loss and health in obesity - An update. Biomed Pharmacother. 2021 Aug;140:111789. doi: 10.1016/j.biopha.2021.111789. Epub 2021 May 31. PMID 34082399
- [Background] Ruban A, Stoenchev K, Ashrafian H, Teare J. Current treatments for obesity. Clin Med (Lond). 2019 May;19(3):205-212. doi: 10.7861/clinmedicine.19-3-205. PMID 31092512
- [Background] De Lorenzo A, Gratteri S, Gualtieri P, Cammarano A, Bertucci P, Di Renzo L. Why primary obesity is a disease? J Transl Med. 2019 May 22;17(1):169. doi: 10.1186/s12967-019-1919-y. PMID 31118060
- [Background] Schetz M, De Jong A, Deane AM, Druml W, Hemelaar P, Pelosi P, Pickkers P, Reintam-Blaser A, Roberts J, Sakr Y, Jaber S. Obesity in the critically ill: a narrative review. Intensive Care Med. 2019 Jun;45(6):757-769. doi: 10.1007/s00134-019-05594-1. Epub 2019 Mar 19. PMID 30888440